CLINICAL TRIAL: NCT03110471
Title: Nurse-led Medicines' Monitoring in Care Homes: a Process Evaluation of the Impact and Sustainability of the West Wales Adverse Drug Reaction (WWADR) Profile and Pharmacist Involvement
Brief Title: Nurse-led Medicines' Monitoring in Care Homes: a Process Evaluation
Status: Completed | Type: Observational
Sponsor: Swansea University (Other)
Collaborators: Abertawe Bro Morgannwg University Health Board (Other)
Responsible Party: Principal Investigator, Professor Sue Jordon, Prof Susan Jordan, Swansea University
Other Study IDs: SwanseaUCHHS
Record Dates: First submitted 2017-03-22; First posted 2017-04-12 (Actual); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Dementia
Keywords: Cognitive impairment; antipsychotics; antidepressants
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Glangarnant Care Home: This is a 'before and after' observational study involving 10 care homes, listed below as groups. The investigators will observe the changes in detection and management of adverse drug reactions between usual care and with administration of the West Wales ADR Profile. Usual care will be provided before and during the intervention period.
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care
- Fieldbay Care Homes: All groups are having identical intervention, so the above text applies to all.
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care
- Neuadd Drymmau Care Home: As above
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care
- Monkstone House,: As above
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care
- Danygraig House: As above
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care
- Ty Coch: As above
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care
- Swn y mor: As above
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care
- Hengoed court: As above
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care
- Hengoed park: As above
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care
- Cefn Lodge care home: As above
  Interventions: Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile; Behavioral: usual care

INTERVENTIONS:
Behavioral: West Wales Adverse Drug Reaction (WWADR) Profile — Nurse-led medicines' monitoring in care homes: a process evaluation of the impact and sustainability of the West Wales Adverse Drug Reaction (WWADR) Profile and pharmacist involvement
Behavioral: usual care — usual care

SUMMARY:
Lay Summary:

The investigators have shown in randomised controlled trials and observation studies that structured nurse-led medicines' monitoring using the WWADR Profile benefits patients, for example, by reducing pain and sedation and identifying high risk cardiovascular conditions. The investigators now aim to understand what is needed to sustain implementation of the WWADR Profile in routine practice and explore future directions.

The participants of the investigators previous research, 5 newly recruited care homes, and stakeholders - care home managers, carers, healthcare professionals, and service users - will be asked to contribute interviews, observations and reflective diaries/ accounts. The investigators are interested in their experiences of medication use, medication management, adverse effects and barriers and facilitators of medicine monitoring, and how electronic devices can enhance nurse-led monitoring.

DETAILED DESCRIPTION:
Background:

Between 1 in 4 and 1 in 25 people benefit from their prescribed medicines (Schork 2015). However, adverse drug reactions (ADRs, known as side effects) occur in 7.8% (7.2-8.4%) patients in community (or ambulatory) care (Hakkarainen et al 2013). Most of these are preventable (Hakkarainen et al 2013, NICE 2015). Adverse drug events (ADE), which include ADRs and under-prescribing, and medicines' mismanagement are responsible for 8% of healthcare spend in the USA, $213bn (Aitkin & Valkova 2013) and 9.5% of direct costs in Sweden.

The West Wales ADR Profiles for medicines' monitoring has improved quality of care by reducing the prescription of mental health medicines and identifying and addressing previously unsuspected adverse effects, such as coupled beats and severe hypertension (Jordan 2002, et al 2002), infections (Gabe el al 2014), chest pain and valproate-induced pancreatitis (Jones et al 2016), and, in care homes, drug-induced Parkinson's (Jordan et al 2014), pain, nausea and behaviour problems (Jordan et al 2015). The investigators now need to know how the intervention can embed in practice and governance frameworks, and benefit from pharmacist involvement and new monitoring devices.

Aims and objectives:

The investigators aim to explore

1. What is needed to sustain implementation of the WWADR Profile in routine practice
2. How it might be enhanced by a) pharmacist involvement and b) digitisation and new monitoring technology c) new profiles in other areas, such as respiratory medicine, pain control, falls.

Research Design A qualitative process evaluation and audit of interest

Duration 9 months from approval date

Location Care homes in Abertawe Bro Morgannwg University Health Board U.K.

The investigators have received full approval from the West Wales Research Ethics Committee,Committee (reference 16/WA/038, IRAS ID 213050), to carry out this study. Written informed consent will be sought for all interviews, observations (service users and nurses), and reviews of reflective diaries or accounts. Copies of the consent forms will be placed in service users' records or given to the interviewees, as appropriate, and stored by the research team in a locked cabinet in a locked office. Participants or their consultees will be free to withdraw or retract their data at any time. Swansea University are the study sponsors and provide indemnity cover.

Recruitment All 5 care homes from the previous trial (Jordan et al 2015) and 5 new care homes have opted to participate.

Methods:

The investigators will use interviews, observations and reflective diaries/ accounts with the participants of 5 previous research sites, and 5 newly recruited care homes.

The investigators propose to explore 2 additions to nurse-led medicines' monitoring:

* Cluster pharmacist or study pharmacist review completed Profiles in a pilot
* Combining administration with the Multiparametric sensor systems (Yang et al 2015) or electronic version of the Profiles in an audit of interest.

Data Handling- All data will be anonymised immediately, and kept strictly confidential. Participants and care homes will be assigned study numbers, and personal names will only appear on consent forms. A file linking care homes' names and addresses to study numbers will be stored in a password protected file on a password protected computer in a locked office used only by the PI. Service users' ages, sex, medicines and medical conditions will be recorded. Professionals' roles and length of service will be recorded. Data will be managed in accordance with the Data Protection Act 1998, the Caldicott Guardian, the Research Governance Framework for Health & Care Research Wales, and the Research Ethics' Committee. Study documents will be stored in locked filing cabinets in a locked office for sole use of the PI. All study data will be anonymised before being entered into electronic files, which will be stored on pass-word protected computers for sole use of the researchers.

Consent- Prospective service user participants will be approached by their nurses. onsent to participation will be obtained by a qualified member of staff who is aware of the Mental Capacity Act 2005. For those without capacity to consent, as this is not a CTIMP, their consultees will be approached for advice regarding involvement. For many participants the consultee is a relative in regular contact; however, some service users have no regular visitors, and rely on professional support. Information sheets (in English and Welsh) and verbal information will be offered and potential participants will be given at least a week to decide whether to be observed or interviewed. Residents (or their family or consultees) to be observed will be asked to sign consent to non-participant observation and review of case notes.

Service users' and carers' views will be obtained as part of this project.

Anticipated outcome: The enhanced Profiles will offer a measure of care quality that matters to service users for example, pain, sedation, food and fluid intake and a sustainable strategy to improve care quality by: a) regular systematic review and transfer of information to pharmacists and prescribers (Francis 2013, Andrews and Butler 2014, Older People's Commissioner 2014, Flynn 2015); b) integration with NHS services e.g. contacts with prescribers, GPs, dentists and opticians; c) pharmacist reviews to optimise medication regimens for participants.

Outcomes to be reported:

Number and nature of problems addressed (including prescription changes)and understanding of any changes needed to optimise clinical gain and sustain implementation.

ELIGIBILITY:
Care Homes.

Inclusion criteria:

Providing residential or nursing care or both to >4 service users meeting inclusion criteria below.

Willing to use the WWADR monitoring Profile in routine practice

Exclusion criteria:

<5 residents meet the inclusion criteria Unwilling or unable to volunteer to undertake nurse-led medicines' monitoring

Inclusion Criteria service users:

* Inclusion criteria:

  * Resident at the care home and expected to continue to be for 1 year;
  * Currently taking one of antipsychotics, anti-epileptics/ mood stabilisers, antidepres-sants, benzodiazepines, Z drugs;
  * Diagnosis of dementia, or dementia related condition, recorded; permanent local authority funding for dementia care; permanent cognitive impairment, but no diagnosis in care home notes.
  * Willing and able to give informed, signed consent themselves, or where capacity is lacking, a consultee who is willing to give advice

Exclusion Criteria:

* • Not well enough to participate, as screened by their nurses;

  * Aged <18;
  * Receiving active palliative care.

Professionals

Inclusion criteria

* Involved in the provision of care for service users described above
* Willing to participate in the study

Exclusion criteria

* Not involved with service users in care homes
* Unwilling to consent to participation

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will work with healthcare professionals and service users involved in care homes in South West Wales.
  The target population for nurse-led medicines' monitoring is care home service users receiving at least one of: antipsychotics, anti-epileptics/ mood stabilisers, antidepressants, anxiolytics or hypnotics (benzodiazepines or Z drugs). Up to 3 service users per care home will be observed. Care homes will be invited to participate in the pilot work with pharmacists.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United Kingdom (10):
  - Llys Gywn Residential Home, Cardiff, Cardiff, Wales
  - Monkstone House, Cardiff, Wales
  - Danygraig House, Cardiff, Wales
  - Neuadddrymmau care home, Swansea, Wales
  - Cefnlodge Care Home, Swansea, Wales
  - Swn-y-mor care home, Swansea, Wales
  - Glangarnant care home, Swansea, Wales
  - Fieldbay Ltd, Swansea, Wales
  - Three Cliffs Care Home, Swansea
  - Glais Care Home, Swansea

IPD SHARING:
Plan to Share IPD: No
Individual participant data, will not be shared & participants not identified. The investigators aim to publish the outcomes in 2018. Swansea university website.

REFERENCES:
- [Background] Schork NJ. Personalized medicine: Time for one-person trials. Nature. 2015 Apr 30;520(7549):609-11. doi: 10.1038/520609a. No abstract available. PMID 25925459
- [Background] Hakkarainen KM, Andersson Sundell K, Petzold M, Hagg S. Prevalence and perceived preventability of self-reported adverse drug events--a population-based survey of 7099 adults. PLoS One. 2013 Sep 4;8(9):e73166. doi: 10.1371/journal.pone.0073166. eCollection 2013. PMID 24023828
- [Background] NICE Medicines and Prescribing Centre (UK). Medicines Optimisation: The Safe and Effective Use of Medicines to Enable the Best Possible Outcomes. Manchester: National Institute for Health and Care Excellence (NICE); 2015 Mar. Available from http://www.ncbi.nlm.nih.gov/books/NBK305021/ PMID 26180890
- [Background] Aitken M. & Valkova S. (2013). Avoidable costs in US Healthcare. IMS Institute for Healthcare Informatics, Parsippany, NJ, USA
- [Background] Jordan S. Managing adverse drug reactions: an orphan task. J Adv Nurs. 2002 Jun;38(5):437-48. doi: 10.1046/j.1365-2648.2002.02205.x. PMID 12028277
- [Background] Jordan S, Tunnicliffe C, Sykes A. Minimizing side-effects: the clinical impact of nurse-administered 'side-effect' checklists. J Adv Nurs. 2002 Jan;37(2):155-65. doi: 10.1046/j.1365-2648.2002.02064.x. PMID 11851783
- [Background] Gabe ME, Murphy F, Davies GA, Russell IT, Jordan S. Medication monitoring in a nurse-led respiratory outpatient clinic: pragmatic randomised trial of the West Wales Adverse Drug Reaction Profile. PLoS One. 2014 May 5;9(5):e96682. doi: 10.1371/journal.pone.0096682. eCollection 2014. PMID 24798210
- [Background] Jones R, Moyle C, Jordan S. Nurse-led medicines monitoring: a study examining the effects of the West Wales Adverse Drug Reaction Profile. Nurs Stand. 2016 Nov 30;31(14):42-53. doi: 10.7748/ns.2016.e10447. PMID 27902153
- [Background] Jordan S, Gabe M, Newson L, Snelgrove S, Panes G, Picek A, Russell IT, Dennis M. Medication monitoring for people with dementia in care homes: the feasibility and clinical impact of nurse-led monitoring. ScientificWorldJournal. 2014 Feb 23;2014:843621. doi: 10.1155/2014/843621. eCollection 2014. PMID 24707218
- [Background] Jordan S, Gabe-Walters ME, Watkins A, Humphreys I, Newson L, Snelgrove S, Dennis MS. Nurse-Led Medicines' Monitoring for Patients with Dementia in Care Homes: A Pragmatic Cohort Stepped Wedge Cluster Randomised Trial. PLoS One. 2015 Oct 13;10(10):e0140203. doi: 10.1371/journal.pone.0140203. eCollection 2015. PMID 26461064
- [Background] Yang S, Chen YC, Nicolini L, Pasupathy P, Sacks J, Su B, Yang R, Sanchez D, Chang YF, Wang P, Schnyer D, Neikirk D, Lu N. "Cut-and-Paste" Manufacture of Multiparametric Epidermal Sensor Systems. Adv Mater. 2015 Nov 4;27(41):6423-30. doi: 10.1002/adma.201502386. Epub 2015 Sep 23. PMID 26398335
- [Background] Francis, R. (2013) Report of the Mid Staffordshire NHS Foundation Trust Public Inquiry. London: The Stationery office. http://www.midstaffspublicinquiry.com/report.
- [Background] Andrews J, Butler M. Trusted to Care: An independent Review of the Princess of Wales Hospital and Neath Port Talbot Hospital at Abertawe Bro Morgannwg University Health Board People, Dementia Services Development Centre, the People Organisation. 2014. Available at: http://wales.gov.uk/docs/dhss/publications/140512trustedtocareen.pdf
- [Background] Flynn M. 2015 In Search of Accountability. Welsh Government, Cardiff, OGL Crown copyright 2015 WG25658 ISBN 978 1 4734 4027 2
- [Background] Older People's Commissioner for Wales. A Place to Call Home. Older people's Commissioner for Wales, Cardiff. 2014. Available at: http://www.olderpeoplewales.com/Libraries/Uploads/A_Place_to_Call_Home_-_A_Review_into_the_Quality_of_Life_and_Care_of_Older_People_living_in_Care_Homes_in_Wales.sflb.ashx
- [Background] Jordan S, Knight J, Pointon D. Monitoring adverse drug reactions: scales, profiles, and checklists. Int Nurs Rev. 2004 Dec;51(4):208-21. doi: 10.1111/j.1466-7657.2004.00251.x. PMID 15530161
- [Background] Jordan S, Banner T, Gabe-Walters M, Mikhail JM, Round J, Snelgrove S, Storey M, Wilson D, Hughes D; Medicines Management Group. Nurse-led medicines' monitoring in care homes study protocol: a process evaluation of the impact and sustainability of the adverse drug reaction (ADRe) profile for mental health medicines. BMJ Open. 2018 Sep 28;8(9):e023377. doi: 10.1136/bmjopen-2018-023377. PMID 30269073
- [Result] Jordan S, Banner T, Gabe-Walters M, Mikhail JM, Panes G, Round J, Snelgrove S, Storey M, Hughes D; Medicines' Management Group, Swansea University. Nurse-led medicines' monitoring in care homes, implementing the Adverse Drug Reaction (ADRe) Profile improvement initiative for mental health medicines: An observational and interview study. PLoS One. 2019 Sep 11;14(9):e0220885. doi: 10.1371/journal.pone.0220885. eCollection 2019. PMID 31509537
- See also: How the west wales adr profiles work — http://www.swansea.ac.uk/adre/
- Available data/document: Publications — http://orcid.org/0000-0002-5691-2987 — Prof Sue Jordan- publication list

RESULTS

PARTICIPANT FLOW:
Groups:
- Observed Residents: The administration of ADRe by nurses with 30 residents was observed in ten volunteer care homes in South West Wales, U.K. Five care homes were recruited to the study from our earlier randomised controlled trial [24], and five were newly recruited. All observed residents were receiving prescribed mental health medicines. The wider policy context was explored in 30 interviews with service users, including family members, nurse managers and strategic health care leads in South Wales
- Service Providers: pharmacists nurses strategic leads
Period: Overall Study
Arm/Group | Observed Residents | Service Providers
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data not collected on the service providers and users.
Groups:
- Observed Residents: Administration of ADRe by nurses to 30 residents in care homes observed
- Service Providers and Users: Policy context explored in interviews with service users, nurse managers strategic leads
- Total: Total of all reporting groups
Arm/Group | Observed Residents | Service Providers and Users | Total
Number analyzed (Participants) | 30 | 0 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 28 | 0 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (9.9) |  | 77.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 |  | 15
  Male | 15 |  | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 |  | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions (ADRs) Treated
Description: ADRs (adverse drug reactions) (as listed in the British National Formulary and manufacturers' datasheets) where actions are taken to correct the problem.
Time Frame: 6 months
Population: Observation of residents. Service providers and users were not observed: they gave interviews.
Measure: Count of Participants; unit: Participants
Groups:
- Whole Study - Observed Residents: Care home (long-stay) residents observed for adverse drug reactions.
Arm/Group | Whole Study - Observed Residents
Number analyzed (Participants) | 30
Participants | 30

2. Secondary Outcome: Time for ADRe Administration (Including Interruptions) in Minutes
Description: Assessed by researchers observing resident/ care-giver interaction.
Time Frame: up to 1 hour
Population: Observed resident/ care-giver interaction.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Whole Study - Observed Residents
Number analyzed (Participants) | 30
minutes | 27.7 (12.0)

3. Secondary Outcome: Number of Problems Identified Per Resident
Description: Signs and symptoms of prescribed medicines as listed as undesirable effects in manufacturers' Summaries of Product Characteristics.
Time Frame: up to 1 hour
Population: Observed resident/ care-giver interaction.
Measure: Mean (Standard Deviation); unit: problems / resident
Arm/Group | Whole Study - Observed Residents
Number analyzed (Participants) | 30
problems / resident | 17.5 (7.1)

4. Secondary Outcome: Number of Changes to Care by Nurses Identified Per Resident
Description: Measures taken to alleviate signs and symptoms of prescribed medicines as listed as undesirable effects in manufacturers' Summaries of Product Characteristics.
Time Frame: up to 4 weeks
Population: Observed resident/ care-giver interaction.
Measure: Mean (Standard Deviation); unit: care changes / resident
Arm/Group | Whole Study - Observed Residents
Number analyzed (Participants) | 30
care changes / resident | 2.3 (1.6)

5. Secondary Outcome: Number of Pharmacist Recommendations for Prescription Review Per Resident
Description: Recommendations to optimise prescription regimens. These included specific points to review or change.
Time Frame: up to 4 weeks
Population: Observed resident/ medicines charts reviewed in conjunction with the ADRe profile.
Measure: Mean (Standard Deviation); unit: recommended changes / resident
Arm/Group | Whole Study - Observed Residents
Number analyzed (Participants) | 30
recommended changes / resident | 3.8 (2.1)

6. Secondary Outcome: Number of Drug Interactions Per Resident
Description: Regimen entered into the BNF drug interactions checker, and number of interactions flagged up were used for this outcome measure.
Time Frame: up to 4 weeks
Population: Observed resident/ medicines charts reviewed.
Measure: Mean (Standard Deviation); unit: drug interactions / resident
Arm/Group | Whole Study - Observed Residents
Number analyzed (Participants) | 30
drug interactions / resident | 6.1 (5.7)

ADVERSE EVENTS:
Time Frame: 7 months study period.No adverse events related to the intervention reported.
Description: non drug trial. Adverse events from using the ADRe Profile were sought from care-givers at the end of the study. No adverse events were reported. Interviewees were not evaluated for adverse events associated with the study.
Groups:
- Observed Residents: This observation study had only one arm (intervention).
Arm/Group | Observed Residents
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT03110471/Prot_000.pdf